CLINICAL TRIAL: NCT00240266
Title: A Randomised, Double-blind, Placebo-controlled, Crossover Pilot Study to Define the High Density Lipoprotein Cholesterol (HDL-C)-Raising Mechanism of Rosuvastatin (CRESTOR™) by Quantifying the Key Steps of Reverse Cholesterol Transport (RCT)
Brief Title: Study of High Density Lipoprotein Cholesterol (HDL-C)-Raising Mechanism of Rosuvastatin (CRESTOR™) by Quantifying the Key Steps of Reverse Cholesterol Transport (RCT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4522AS/0003
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Metabolic Syndrome; Dyslipidemia
Keywords: Metabolic Syndrome; Dyslipaemia
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor

SUMMARY:
The purpose of this study is to investigate the effect of treatment with rosuvastatin on the capacity of plasma to promote cholesterol efflux, which is the first and likely rate limiting step in reverse cholesterol transport.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* males aged 45-65
* insulin resistance
* central obesity
* LDL-C <6 mmol/L
* plasma triglycerides >=1.7 and ≤5.5 mmol/L
* HDL-C ≤1.2 mmol/L.

Exclusion Criteria:

* total cholesterol >7mmol/L
* pre-existing cardiovascular disease, diabetes, proteinuria or renal failure

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2003-08; Primary Completion 2004-11 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Determine the effect of treatment with rosuvastatin on the capacity of plasma to promote cholesterol efflux, which is the first and likely rate limiting step in reverse cholesterol transport.

SECONDARY OUTCOMES:
Determine the effect of treatment with rosuvastatin on:
- cholesterol esterification by measuring plasma lecithin:cholesterol acyl transferase concentration and capacity to esterify cholesterol, one of the stops in RCT.
- plasma concentration of cholesterol ester transfer protein and capacity to transfer cholesterol from HDL-C to apoB-containing lipoproteins, one of the steps in RCT.
- plasma concentration of preβ1-HDL.
- plasma concentration of LDL cholesterol, HDL-C and apoA-1.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Nestel, MD, Principal Investigator — Baker Heart Research Institute
Locations (1):
- Research Site, Melbourne, Victoria, Australia